CLINICAL TRIAL: NCT03214263
Title: Identification of New Biomarkers to Improve Diagnostics or Predict Treatment Responses, Adverse Events or Prognosis in Patients With Inflammatory Rheumatic Disease Followed in the Danish Nationwide Quality Registry, DANBIO
Brief Title: Identification of New Biomarkers to Promote Personalized Treatment of Patients With Inflammatory Rheumatic Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Copenhagen University Hospital at Herlev (Other); King Christian X´Hospital for Rheumatic Diseases (Other); Svendborg Hospital (Other); Zealand University Hospital (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other); Sygehus Lillebaelt (Other); Odense University Hospital (Other); Hillerod Hospital, Denmark (Other); Randers Regional Hospital (Other); University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Merete L Hetland, Professor, Rigshospitalet, Denmark
Other Study IDs: REUM BIOMARKØRER 2014-10-30
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Arthritis, Rheumatoid; Psoriatic Arthritis; Axial Spondyloarthritis; Connective Tissue Diseases; Gout
Keywords: Inflammatory rheumatic diseases; Biomarkers; Tailored treatment; Personalised medicine; DANBIO; Danish Rheumatologic Biobank; clinical data
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Axial Spondyloarthritis; Connective Tissue Diseases; Gout

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — EDTA-whole blood, EDTA-plasma, EDTA-buffy coat, serum, synovial fluid, tissue, PAXgene RNA tubes
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cross-sectional samples:: Any patient followed in the DANBIO registry may be invited to participate when they meet for a scheduled routine clinical visit. These patients provide one cross-sectional blood sample.
- Longitudinal samples:: Any patient followed in the DANBIO registry will be invited to participate when they start treatment with a new DMARD. Switching from csDMARD to bDMARD, or from one bDMARD to another bDMARD indicates a new baseline.
- Samples of other biological material:: Patients followed in the DANBIO registry may be invited to participate if scheduled for one of the following procedures: joint puncture with extraction of synovial fluid, surgery or tissue sampling involving synovia, cartilage, bone, bone-marrow or other tissues. Representative samples from the synovial fluid or relevant tissue are collected after routine diagnostic or therapeutic analyses have been done

SUMMARY:
Introduction: The medical treatment of inflammatory rheumatic diseases has improved dramatically during the last decades primarily due to the introduction of biological disease modifying anti-rheumatic drugs (bDMARDs). However, bDMARD treatment failure occurs in 30-40% of patients due to lack of effectiveness or side effects. The tools to predict treatment outcomes in the individual patient are currently limited. The objective of the present study is to identify diagnostic, prognostic and predictive biomarkers, which can be used to 1) diagnose inflammatory rheumatic diseases early in the disease course with high specificity and sensitivity, 2) improve prognostication or 3) predict treatment effectiveness and tolerability for the individual patient.

Methods and analysis: Observational and translational open cohort study with prospective collection of clinical data and biological materials in patients with inflammatory rheumatic diseases treated in routine care. Patients contribute one cross-sectional blood sample (i.e. whole blood, serum, EDTA-plasma and -buffy coat, and blood in PAXgene RNA tubes) and/or are enrolled for longitudinal follow-up upon start of new DMARD (blood sampling after 0/3/6/12/24/36/48/60 months' treatment). Demographics, disease characteristics, comorbidities and lifestyle factors are registered at inclusion; DMARD treatment and outcomes are collected repeatedly during follow-up. Currently (June 2017) >5,000 samples from ≈3,000 patients have been collected. Data will be analysed using appropriate statistical analyses.

Ethics and dissemination: The protocol is approved by the Danish Ethics Committee and The Danish Data Protection Agency. All participants give written informed consent. Biomarkers will be evaluated and published according to REMARK, STROBE and STARD guidelines. Results will be published in peer-reviewed medical journals and presented at international conferences.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with or suspected for the following diseases: rheumatoid arthritis (RA), psoriatic arthritis (PsA), axial spondyloarthritis (axSpA) or other inflammatory rheumatic diseases, connective tissue disorders or gout
* Aged 18 year or older
* Able to give informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are eligible for inclusion if they are followed in routine care and monitored in DANBIO with one of the following diagnoses: RA, axSpA (including ankylosing spondylitis), PsA, other inflammatory rheumatic diseases, connective tissue disorders or gout, or are suspected for one of the above. Patients must be able to give written informed consent and aged ≥18 years.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2015-05; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To diagnose inflammatory rheumatic diseases early in the disease course with high specificity and sensitivity | Changes from baseline to 3, 6, 12, 24, 36, 48, and 60 months
  Number of patients suspected of rheumatoid arthritis, axial spondyloarthritis, psoriatic arthritis, gout or connective tissue diseases that can be correctly diagnosed
To improve prognostication | At diagnosis and after 3, 6, 12, 24, 36, 48 and 60 months
  Number of patients that can be correctly prognosticated by progression in physical function (by HAQ) and in bone damage (by imaging)
To predict treatment effectiveness and tolerability for the individual patient | At treatment onset and at 3, 6, 12, 24, 36, 48 and 60 months
  Number of patients that achieve a standardized treatment response and do not experience serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Merete L Hetland, Professor, Principal Investigator — Rigshospitalet, Glostrup, Denmark
Locations (11):
- Denmark (11):
  - Department of Rheumatology, Aalborg University Hospital, Aalborg
  - Department of Rheumatology, Aarhus University Hospital, Aarhus
  - Department of Rheumatology, Rigshospitalet, Copenhagen
  - Dept. of Rheumaology, University Hospital Bispebjerg and Frederiksberg, Copenhagen
  - Dept. of Rheumaology, North Denmark Regional Hospital, Hjørring
  - Department of Rheumatology, Zealand University Hospital Køge, Køge
  - Department of Rheumatology, Odense University Hospital, Odense
  - Dept. of Rheumaology, Randers Regional Hospital, Randers
  - Department of Rheumatology, Svendborg Hospital, Svendborg
  - Danish Arthritis Hospital, Sønderborg
  - Department of Rheumatology, Hospital Lillebaelt, Vejle

REFERENCES:
- [Derived] Kringelbach TM, Glintborg B, Hogdall EV, Johansen JS, Hetland ML; Biomarker Protocol Study Group. Identification of new biomarkers to promote personalised treatment of patients with inflammatory rheumatic disease: protocol for an open cohort study. BMJ Open. 2018 Feb 1;8(2):e019325. doi: 10.1136/bmjopen-2017-019325. PMID 29391382
- See also: Bio- and GenomeBank Denmark and Danish Rheumatologic Biobank — http://www.regioner.dk/rbgb
- See also: DANBIO — http://danbio-online.dk/